CLINICAL TRIAL: NCT00840060
Title: AMALS: Addressing Multiple Aspects of Language Simultaneously: A Randomized Clinical Trial
Brief Title: Efficacy of AMALS in Treating Language Impairment in Children
Acronym: AMALS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lamar University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Monica L. Harn, Associate Professor, Speech and Hearing Services, Lamar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RDC009027A-01A2; 1R15DC009027-01A2 (NIH); NIDCD RDC009027A-01A2
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Results first posted 2012-05-15 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Language Disorder
MeSH Terms: conditions — Language Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AMALS (Experimental): Addressing multiple aspects of language simultaneously
  Interventions: Behavioral: AMALS
- DTA (Experimental): Discrete Trial Approach
  Interventions: Behavioral: DTA

INTERVENTIONS:
Behavioral: AMALS — Addressing multiple aspects of language simultaneously
  Arms: AMALS
Behavioral: DTA — Discrete Trial Approach
  Arms: DTA

SUMMARY:
The goal of this proposal is to examine the efficacy of a manualized treatment intervention, AMALS: Addressing Multiple Aspects of Language Simultaneously, which is designed to remediate semantic, morphological, and syntactic aspects of language in preschool children with language impairment. This study will target preschool children with language impairment living in a region characterized by nonmainstream dialects.

Questions driving this work are:

1. Will children participating in the AMALS treatment exhibit greater semantic, morphological, and syntactic complexity on multiple outcome measures at the completion of the intervention compared to a Discrete Trial Approach (DTA) group?
2. Will these gains be maintained at one-month follow up?
3. What is the impact of dialect on dependent variables, specifically morphosyntactic abilities?

To answer these questions a randomized clinical trial will be conducted comparing AMALS, an integrated approach to treatment, with DTA, an additive approach to therapy. In this study rather than restrict the ethnic and cultural backgrounds of this population, children's use of dialect will be uniquely identified and examined.

ELIGIBILITY:
Inclusion Criteria:

1. Demonstrate sufficient intelligibility as determined by a score of 85% on percent consonant correct (PCC) measures;
2. Demonstrate sufficient phonological ability to use grammatical morphemes as determined by use of word-final /s, z, t, d/ on sound- in-word subtest from the Goldman-Fristoe Test of Articulation-2 (GFTA; Goldman & Fristoe, 2000)
3. Nonverbal IQ above 70 as scored on the Columbia Mental Maturity Scale (CMMS; Burgemeister, Blum, & Lorge, 1972);
4. Below 1SD on the Diagnostic Evaluation of Language Variation: Norm-referenced Test (DELV; Seymour, Roeper & de Villiers, 2005);
5. Below 1.39SD on the Structured Photographic Expressive Language Test-Preschool (SPELT-P; Werner & Kresheck, 1983);
6. Documentation from teachers and/or parents of impressions of language status in comparison with peers;
7. More than one standard deviation below the mean on both levels 3 and 4 of the Preschool Language Assessment Instrument (PLAI; Blank, Rose, & Berlin, 1978).

Exclusion Criteria:

1. English as the primary language
2. No oral-motor impairment
3. No hearing impairment
4. No co-morbid psychiatric or neurological impairments

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica L Bellon-Harn, Ph.D., Principal Investigator — Lamar University
Locations (3):
- United States (3):
  - West Orange Cove Consolidated Independent School District, Orange, Texas
  - Little-Cypress Mauriceville Consolidated School District, Orange, Texas
  - Port Arthur Independent School District, Port Arthur, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children were recruited at three public school sites. From January 2009 to May 2010, 50 participants were successfully recruited. Of the 50, 40 met inclusion criteria and were randomly assigned to one of the two treatments.
Pre-assignment Details: No participants were excluded from the treatment following enrollment.
Groups:
- Addressing Multiple Aspects of Language Simultaneously: Children assigned to this treatment group participated in language treatment that followed a scaffolded-language structure. Linguistic content and structures were not explicitly targeted.
- Discrete Trial Approach: Children assigned to this treatment group participated in a language treatment following an additive structure. Linguistic content and structure were explicitly targeted.
Period: Overall Study
Arm/Group | Addressing Multiple Aspects of Language Simultaneously | Discrete Trial Approach
Started | 20 | 20
Completed | 19 | 19
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Change in emotional/behavioral status | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Addressing Multiple Aspects of Language Simultaneously | Discrete Trial Approach | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 20 | 40
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 4.56 (.50) | 4.90 (.51) | 4.74 (.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 11 | 14 | 25
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Language Sample Analysis
Description: Samples were transcribed and segmented by utterance. Each was coded categorically. Reported measures include percentage of utterances at the interpretive/inferential label, percentage of utterances with one or more t-unit (i.e., noun phrase + verb phrase), percentage of utterances that required copula (is/are) or auxiliary (is/are) that were produced.
Time Frame: Language samples were obtained pre-treatment, post-treatment, and at one-month follow-up.
Population: Language samples were collected for all children participating in either treatment condition.
Measure: Mean (Standard Deviation); unit: Percentage of utterances
Arm/Group | Addressing Multiple Aspects of Language Simultaneously | Discrete Trial Approach
Number analyzed (Participants) | 19 | 19
Percentage of utterances
  Interpretive utterances: pre-treatment | 17.33 (3.31) | 18.00 (3.22)
  Interpretive utterances: post-treatment | 39.35 (4.04) | 26.38 (3.92)
  Interpretive utterances: 1-month follow-up | 39.70 (4.16) | 20.55 (4.04)
  T-units: pre-treatment | 52.30 (21.00) | 53.77 (22.70)
  T-units: post-treatment | 80.94 (13.18) | 69.78 (20.19)
  T-units: one-month follow-up | 74.88 (16.99) | 55.83 (29.48)
  Frequency of copula (is/are): pre-treatment | 56.00 (33.24) | 71.00 (33.59)
  Frequency of copula (is/are): post-treatment | 77.05 (26.78) | 76.43 (26.12)
  Frequency of copula (is/are): 1-month follow-up | 76.94 (25.72) | 75.81 (23.55)
  Frequency of auxiliary (is/are): pre-treatment | 40.11 (38.87) | 48.87 (35.13)
  Frequency of auxiliary (is/are): post-treatment | 65.23 (23.73) | 59.12 (26.02)
  Frequency of auxiliary (is/are): 1-month follow-up | 50.23 (34.15) | 48.68 (24.51)

2. Primary Outcome: Number of Verb Structures Per Utterance
Description: Samples were transcribed and segmented by utterance. Utterances were analyzed for novel verb structures. Structures were included if they were produced more than one time.
Time Frame: Pre-treatment, post-treatment, 1-month follow-up
Measure: Mean (Standard Deviation); unit: Novel verb structures per utterance
Arm/Group | Addressing Multiple Aspects of Language Simultaneously | Discrete Trial Approach
Number analyzed (Participants) | 19 | 19
Novel verb structures per utterance
  Novel verb structures per utterance: pre-treatment | 3.52 (2.26) | 4.15 (2.16)
  Novel verb structure per utterance: post-treatment | 5.94 (1.59) | 4.61 (1.78)
  Novel verb structures per utterance: 1-month follo | 5.41 (2.78) | 4.16 (2.20)

ADVERSE EVENTS:
Arm/Group | Addressing Multiple Aspects of Language Simultaneously | Discrete Trial Approach
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
Problems with stratification according to dialect prior to randomization lead to difficulty interpreting results related to dialect

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes